CLINICAL TRIAL: NCT05258617
Title: Low-Level Laser Therapy Treatment of Lung Inflammation in Post-COVID-19 Recovery
Status: Terminated | Type: Observational
Why Stopped: Study was associated with a declining population - COVID 19. Difficulty recruiting participants.
Sponsor: Ward Photonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CP21-01
Record Dates: First submitted 2022-02-24; First posted 2022-02-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: LLLT Photobiomodulation — Treatment with red LED light using UltraSlim device.

SUMMARY:
An informational evaluation of COVID-19 patients who receive low-level laser therapy in addition to a normal regimen of treatment for symptoms associate with COVID-19. Results are compared to statistical observations published in literature from patients receiving standard care for COVID-19 symptoms without low-level laser therapy.

DETAILED DESCRIPTION:
Since the emergence of COVID-19, the world has become familiar with the symptoms and acute effects of COVID-19 infection including hospitalization and death. However, we now know that COVID-19 can cause persistent ill-health even after patients recover from active infection. Around a quarter of people who have had the virus experience symptoms that continue for at least a month but one in 10 are still unwell after 12 weeks. This has been described by patient groups as "Long COVID," a colloquial term used to describe signs and symptoms that continue or develop after the acute phase of the coronavirus (COVID-19). This encompasses the terms "ongoing symptomatic COVID-19" (4 to 12 weeks after infection) and "post-COVID-19 syndrome" (more than 12 weeks after infection).

Data from recent studies shows that approximately 9-15% of patients who were hospitalized with COVID-19 are readmitted within two months of discharge, and nearly 30% are readmitted within six months of discharge.

This highlights the fact that sequelae after recovery from acute COVID19 may require ongoing treatment to help return patients to their prior quality of life. Reasons for hospital readmission in these post-covid recovery patients range from respiratory distress, sepsis, pneumonia, heart failure, thrombotic episodes, psychiatric illness, and falls, among other causes. Risk factors for readmission have included older age, certain underlying conditions (e.g., chronic obstructive pulmonary disease, hypertension), shorter initial length of stay, and lower rates of in-hospital treatment-dose anticoagulation

The prevalence of long COVID symptoms and accompanying respiratory inflammation are understood through statistical survey of populations. A study conducted by the MICOVID19 (Michigan) initiative in July 2020 documented post-COVID recovery rates of 1,648 patients. The goals of the Michigan registry are to Identify factors associated with critical illness/severe course and outcomes, Identify patient characteristics, care practices, and treatment regimens associated with improved outcomes, and Understand the long-term complications for hospitalized patients including subsequent rates of readmission, mortality, and return-to-normal activities (among other specific state goals).Post-acute COVID-19 is defined as persistent symptoms and/or delayed or long-term complications after having moved through the acute phase of the illness.

The MICOVID19 study will serve as a standard comparison to the results of this study, and will show whether patients treated with LLLT red light using the UltraSlim device have statistically better outcomes than the patients surveyed in the MICOVID19 study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is diagnosed with COVID-19
* Study participant is 18 years of age or older
* Patient exhibiting moderate-to-acute respiratory distress

Exclusion Criteria:

* Photosensitive condition or medication
* Active chemotherapy treatment or other cancer treatment
* Autoimmune Disorder
* Pregnant, possibly pregnant or planning pregnancy prior to the end of study participation
* Under 18
* Active cancer
* pre-existing pulmonary disease (asthma chronic bronchitis, emphasema
* Developmental disability or cognitive impairment that, in the opinion of the investigator, would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have been infected with COVID-19, but no longer active virus, and who have lingering acute respiratory effects from infection.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Decreased inflammation of the lungs | 3 weeks
  Inflammation of the lungs is decreased more for patients treated with LLLT in addition to the standard treatments for COVID-19 than patients who do not receive LLLT treatments as compared to literature studies available for comparison. The decrease in inflammation is measured by showing statistical improvements in O2 saturation, D-Dimer levels, C-reactive Protein, and IL-6 levels.

SECONDARY OUTCOMES:
Subjective assessment of overall health | 3 weeks
  A secondary objective of the trial is to determine whether quality of life/well-being is improved for patients suffering from lingering health effects from COVID-19 by using LLLT treatment post-COVID. Patient quality of life is improved as measured through subjective assessment (survey) of wellbeing.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - MD at Bedside, Berkeley, California
  - Health Atlast, Los Angeles, California
  - Longevity, Santa Monica, California
  - Wellness Junction, Millsboro, Delaware
  - Diet MD, Honolulu, Hawaii
  - Diet MD, ‘Ewa Beach, Hawaii
  - Healing Health Services, Brooklyn, New York